CLINICAL TRIAL: NCT01239472
Title: Cytokines Evaluation in Early Calcineurin Inhibitors Withdrawn on Renal Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andre Barreto Pereira (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Andre Barreto Pereira, MD, Msc, PhD, Santa Casa de Misericórdia de Belo Horizonte
Organization: Santa Casa de Misericórdia de Belo Horizonte (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001ABR14T
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Renal Transplant Rejection; Immunosuppression
Keywords: chronic allograft nephropathy; cytokines; kidney transplant; calcineurin inhibitors withdrawn
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tacrolimus (No Intervention): Kidney transplant patients with living or deceased donors using tacrolimus, mycophenolate sodium and prednisone.
- everolimus (Active Comparator): Kidney transplant patients with living or deceased donors using tacrolimus, mycophenolate sodium and prednisone, and converted for everolimus, mycophenolate sodium, and prednisone 90 days after renal transplantation.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Replacement of tacrolimus by everolimus, 30 days after transplat. It was done after kidney biopsy (excluding acute rejection), blood and urine analysis.
  Other Names: Certican
  Arms: everolimus

SUMMARY:
Currently, acute kidney injury is diagnosed by increased serum creatinine. However, creatinine is not a reliable marker for acute changes in renal function.

The biology of the renal graft is influenced by chemokines from reperfusion (just after the kidney transplant) and throughout its course, when acute and chronic inflammatory changes occurs. Moreover, the evaluation of changes in urinary cytokines reflects kidney interstitial patterns, and can predict renal function, acute rejection episodes and their response to treatment.

Today there are several studies comparing the relative immunosuppression of renal function, but few noticed its relationship with cytokines and chemokines. Thus, we proposed studying the inflammatory consequences of early calcineurin inhibitors (ICN) withdrawing in transplant patients by urine analysis. Kidney biopsy was done before ICN withdrawn and replaced by everolimus (3 months after transplant), and 1 year after transplant.

DETAILED DESCRIPTION:
1. Research objectives

   OBJECTIVES

   Main Objectives:

   • Evaluate the urinary chemokines in kidney transplant patients taking prednisone, tacrolimus and mycophenolate sodium compared to those in use prednisone, mycophenolate sodium and everolimus as maintenance immunosuppression.

   Secondary Objectives:

   • Assess renal function (serum creatinine and its clearance estimated by the Cockcroft-Gault) and a composite outcome (acute rejection, graft loss, death and abandonment of the study) in patients taking prednisone, tacrolimus and mycophenolate sodium compared to those taking prednisone, mycophenolate sodium and everolimus as maintenance immunosuppression.
2. Scientific background, relevance and justification of the research

In current clinical practice, acute kidney injury is typically diagnosed by measuring serum creatinine. Unfortunately, creatinine is an unreliable indicator during acute changes in kidney function. First, serum creatinine concentrations may not change until about 50% of kidney function has already been lost. Second, serum creatinine does not accurately depict kidney function until a steady state has been reached, which may require several days. Chemokines can influence at least three aspects of the biology of the renal graft: 1 - the restoration of blood flow in the graft can lead to injury type ischemia / reperfusion in which chemokines recruit leukocytes; 2 - receptor responses to infection during immune suppression involve chemokines and 3 - the inflammatory components in the acute rejection (RA) and interstitial fibrosis / tubular atrophy (IF/TA) are controlled by chemokines.

Current data have showed urinary cytokines predicting renal function by months in renal transplanted patients. In the evaluation of urinary cytokines and chemokines in the presence of acute rejection, taken together the studies reported elevations of urinary levels of Protein-3 alpha (MIP-3α/CCL20), interleuxin-8 (IL-8/CXCL8), interleuxin-6 (IL-6), tumoral necrosis factor (TNF), interleukin- 10 (IP-10), interferon (IFN), monocyte chemoattractant protein-1 (MCP-1 / CCL2), Interferon gamma-induced protein 10 (IL-10), Monokine induced by gamma interferon (MIG/CXCL9), Interferon-inducible T-cell alpha chemoattractant (I-TAC/CXCL11), regulated upon activation normal T cell expressed and secreted (RANTES/CCL5). As predictors of complications and future changes in renal function, levels of Transforming growth factor beta (TGF-β) and interferon-gamma inducible protein 10 (IP-10/CXCL10) were associated with renal function 6 months and 4 years after transplantation (15-16). IP-10/CXCL10, MIG/CXCL9, G protein-coupled receptor 9 (GPR9/CXCR3), RANTES/CCL5 and the percentage of binding of interleukin-2 (IL-2) were associated with the occurrence of RA. IP-10/CXCL10 and MIG/CXCL9 were also considered useful as predictors of response to treatment of RA. Nankivell et al reported in 2003 that after 1year of renal transplant, 94% of patients present with chronic rejection grade I (BANFF score) and 76% present with calcineurin nephrotoxicity, although there is insufficient data about urinary cytokines at these situations. And adding new information, Hu et al reported in 2009 urinary major intrinsic protein-delta (MIP-δ), osteoprotegerin (OPG), IP-10/CXCL10, MIG/CXCL9 as good biomarkers for acute renal rejection and IF/TA.

Nowadays there is a lot of studies comparing immunosuppression in relation to renal function but not so much in relation to chemokines and cytokines, which are more representative of allograft inflammation and fibrosis.

So, we proposed studying the inflammatory consequences of early CNI withdrawn in renal transplant patients before the immunosuppression modification (3 months after transplant) and 1 year after kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old and under 65 years old
* Recipients of first kidney transplant
* Donor younger than 65 years old
* PRA (panel reactive antigen) ≤ 30% in class I or class II
* No acute rejection episodes
* Proteinuria <1000 mg / day

Exclusion Criteria:

* multiple organ transplant recipient
* Chronic liver failure
* Asymptomatic bacteriuria or urinary infection at randomization time
* Creatinine ≥ 2 mg / dL at randomization time (90 days after transplant)
* Presence of uncontrolled hypercholesterolemia (≥ 350 mg / dL, ≥ 9.1 mmol / L) or hypertriglyceridemia (≥ 500 mg / dL, ≥ 5.6 mmol / L) at randomization time (90 days after transplant)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre B Pereira, PhD, Principal Investigator — Marieta Konder Bornhausen Hospital and Maternity
Locations (1):
- Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared in this website, and in the publication that is already being written.
Supporting Information: Study Protocol, SAP
Time Frame: Data are already available in this website, and will keep available with the PI for 1 year after the publication.
Access Criteria: All data will be available in this website and with the PI, Dr Andre Barreto Pereira, by his e-mail.

REFERENCES:
- [Background] Devarajan P. Emerging biomarkers of acute kidney injury. Contrib Nephrol. 2007;156:203-12. doi: 10.1159/000102085. PMID 17464129
- [Background] Hu H, Knechtle SJ. Elevation of multiple cytokines/chemokines in urine of human renal transplant recipients with acute and chronic injuries: potential usage for diagnosis and monitoring. Transpl Rev 2006;20:165-71
- [Background] Ruster M, Sperschneider H, Funfstuck R, Stein G, Grone HJ. Differential expression of beta-chemokines MCP-1 and RANTES and their receptors CCR1, CCR2, CCR5 in acute rejection and chronic allograft nephropathy of human renal allografts. Clin Nephrol. 2004 Jan;61(1):30-9. doi: 10.5414/cnp61030. PMID 14964455
- [Background] Sibbring JS, Sharma A, McDicken IW, Sells RA, Christmas SE. Localization of C-X-C and C-C chemokines to renal tubular epithelial cells in human kidney transplants is not confined to acute cellular rejection. Transpl Immunol. 1998 Dec;6(4):203-8. doi: 10.1016/s0966-3274(98)80009-9. PMID 10342733
- [Background] Di Paolo S, Gesualdo L, Stallone G, Ranieri E, Schena FP. Renal expression and urinary concentration of EGF and IL-6 in acutely dysfunctioning kidney transplanted patients. Nephrol Dial Transplant. 1997 Dec;12(12):2687-93. doi: 10.1093/ndt/12.12.2687. PMID 9430873
- [Background] Smith SD, Wheeler MA, Lorber MI, Weiss RM. Temporal changes of cytokines and nitric oxide products in urine from renal transplant patients. Kidney Int. 2000 Aug;58(2):829-37. doi: 10.1046/j.1523-1755.2000.00232.x. PMID 10916108
- [Background] Jimenez R, Ramirez R, Carracedo J, Aguera M, Navarro D, Santamaria R, Perez R, Del Castillo D, Aljama P. Cytometric bead array (CBA) for the measurement of cytokines in urine and plasma of patients undergoing renal rejection. Cytokine. 2005 Oct 7;32(1):45-50. doi: 10.1016/j.cyto.2005.07.009. PMID 16153856
- [Background] Prodjosudjadi W, Daha MR, Gerritsma JS, Florijn KW, Barendregt JN, Bruijn JA, van der Woude FJ, van Es LA. Increased urinary excretion of monocyte chemoattractant protein-1 during acute renal allograft rejection. Nephrol Dial Transplant. 1996 Jun;11(6):1096-103. PMID 8671975
- [Background] Grandaliano G, Gesualdo L, Ranieri E, Monno R, Stallone G, Schena FP. Monocyte chemotactic peptide-1 expression and monocyte infiltration in acute renal transplant rejection. Transplantation. 1997 Feb 15;63(3):414-20. doi: 10.1097/00007890-199702150-00015. PMID 9039933
- [Background] Hu H, Aizenstein BD, Puchalski A, Burmania JA, Hamawy MM, Knechtle SJ. Elevation of CXCR3-binding chemokines in urine indicates acute renal-allograft dysfunction. Am J Transplant. 2004 Mar;4(3):432-7. doi: 10.1111/j.1600-6143.2004.00354.x. PMID 14961998
- [Background] Kanmaz T, Feng P, Torrealba J, Kwun J, Fechner JH, Schultz JM, Dong Y, Kim HT, Dar W, Hamawy MM, Knechtle SJ, Hu H. Surveillance of acute rejection in baboon renal transplantation by elevation of interferon-gamma inducible protein-10 and monokine induced by interferon-gamma in urine. Transplantation. 2004 Oct 15;78(7):1002-7. doi: 10.1097/01.tp.0000134397.55564.71. PMID 15480165
- [Background] Hauser IA, Spiegler S, Kiss E, Gauer S, Sichler O, Scheuermann EH, Ackermann H, Pfeilschifter JM, Geiger H, Grone HJ, Radeke HH. Prediction of acute renal allograft rejection by urinary monokine induced by IFN-gamma (MIG). J Am Soc Nephrol. 2005 Jun;16(6):1849-58. doi: 10.1681/ASN.2004100836. Epub 2005 Apr 27. PMID 15857922
- [Background] Kotsch K, Mashreghi MF, Bold G, Tretow P, Beyer J, Matz M, Hoerstrup J, Pratschke J, Ding R, Suthanthiran M, Volk HD, Reinke P. Enhanced granulysin mRNA expression in urinary sediment in early and delayed acute renal allograft rejection. Transplantation. 2004 Jun 27;77(12):1866-75. doi: 10.1097/01.tp.0000131157.19937.3f. PMID 15223905
- [Background] Sorrentino S, Landmesser U. Nonlipid-lowering effects of statins. Curr Treat Options Cardiovasc Med. 2005 Dec;7(6):459-66. doi: 10.1007/s11936-005-0031-1. PMID 16283973
- [Background] Yamada K, Hatakeyama E, Arita S, Sakamoto K, Kashiwabara H, Hamaguchi K. Prediction of chronic renal allograft dysfunction from evaluations of TGFBeta1 and the renin-angiotensin system. Clin Exp Nephrol. 2003 Sep;7(3):238-42. doi: 10.1007/s10157-003-0237-z. PMID 14586721
- [Background] Teppo AM, Honkanen E, Finne P, Tornroth T, Gronhagen-Riska C. Increased urinary excretion of alpha1-microglobulin at 6 months after transplantation is associated with urinary excretion of transforming growth factor-beta1 and indicates poor long-term renal outcome. Transplantation. 2004 Sep 15;78(5):719-24. doi: 10.1097/01.tp.0000131816.51366.6b. PMID 15371675
- [Background] Tatapudi RR, Muthukumar T, Dadhania D, Ding R, Li B, Sharma VK, Lozada-Pastorio E, Seetharamu N, Hartono C, Serur D, Seshan SV, Kapur S, Hancock WW, Suthanthiran M. Noninvasive detection of renal allograft inflammation by measurements of mRNA for IP-10 and CXCR3 in urine. Kidney Int. 2004 Jun;65(6):2390-7. doi: 10.1111/j.1523-1755.2004.00663.x. PMID 15149352
- [Background] Nankivell BJ, Borrows RJ, Fung CL, O'Connell PJ, Allen RD, Chapman JR. The natural history of chronic allograft nephropathy. N Engl J Med. 2003 Dec 11;349(24):2326-33. doi: 10.1056/NEJMoa020009. PMID 14668458
- [Background] Hu H, Kwun J, Aizenstein BD, Knechtle SJ. Noninvasive detection of acute and chronic injuries in human renal transplant by elevation of multiple cytokines/chemokines in urine. Transplantation. 2009 Jun 27;87(12):1814-20. doi: 10.1097/TP.0b013e3181a66b3e. PMID 19543058

RESULTS

PARTICIPANT FLOW:
Groups:
- Tacrolimus: Kidney transplant patients taking tacrolimus, mycophenolate sodium and prednisone the whole study
- Everolimus: Kidney transplant patients taking tacrolimus, mycophenolate sodium and prednisone, whom switched tacrolimus to everolimus 90 days after renal transplantation. Since then the patients kept taking everolimus, mycophenolate sodium and prednisone
Period: Overall Study
Arm/Group | Tacrolimus | Everolimus
Started | 15 | 15
Completed | 10 | 12
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Urine and biopsy data are collected 90 days and 365 days after transplant. Other clinical data as Creatinine, patient information were collected monthly until 365 days after transplant. Among 22 patients included in the study, some urine were lost and couldn't therefore be analysed
Groups:
- Tacrolimus: Kidney transplant patients taking tacrolimus, mycophenolate sodium and prednisone with low immunologic risk .
- Everolimus: Kidney transplant patients taking tacrolimus, mycophenolate sodium and prednisone with low immunologic risk, and converted for use of mycophenolate sodium, everolimus, and prednisone after 90 days of kidney transplantation.
- Total: Total of all reporting groups
Arm/Group | Tacrolimus | Everolimus | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Brazil | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cytokines Evaluation
Description: Cd106(VCAM-1) , IP-10/CXCL10, MIG/CXCL9, MCP-1/CCL2, IL-1, RANTES, IL-8, IL12p70, TNF, IL-10, IL-6, IL-1, VEGF, FGF, CD54(ICAM-1) were analysed in urine 90 days after transplant (before randomization), and 365 days after transplant. Material were conserved at -80 Celsius, and analysed by ELISA at same time. Data was shown in MFI units
Time Frame: Urine and biopsy data are collected 90 days and 365 days after transplant.
Population: 15 patients were enrolled in each group. However in "tacrolimus" group 5 patients didn't want to be submitted to other biopsy and to collect urine 365 days after transplant. And in "everolimus" group 3 patients had adverse events and was switched back to tacrolimus.
Measure: Median (Inter-Quartile Range); unit: MFI
Groups:
- Tacrolimus: Kidney transplant patients taking tacrolimus, mycophenolate sodium and prednisone, during the whole study. This is the no intervention group.
- Everolimus: Kidney transplant patients taking tacrolimus, mycophenolate sodium and prednisone at beginning, but whom switched tacrolimus to everolimus at 90 days after transplant. This is the intervention group
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 10 | 12
MFI
  IP10 90days | 380 [261 to 900] | 893 [194 to 1825]
  IP10 365days | 763 [88 to 1668] | 147 [127 to 353]
  MCP1 90days | 2349 [1751 to 3234] | 4119 [2652 to 7529]
  MCP1 365days | 1306 [750 to 7259] | 1375 [790 to 3342]
  MIG 90days | 396 [239 to 673] | 433 [249 to 1925]
  MIG 365days | 287 [153 to 964] | 580 [262 to 1090]
  RANTES 90days | 148 [134 to 167] | 145 [134 to 212]
  RANTES 365days | 144 [134 to 199] | 155 [151 to 165]
  IL8 90days | 495 [328 to 804] | 624 [409 to 1019]
  IL8 365days | 641 [327 to 1874] | 435 [321 to 558]
  IL12 90days | 116 [110 to 121] | 124 [111 to 130]
  IL12 365days | 124 [119 to 133] | 124 [119 to 138]
  TNF 90days | 136 [134 to 145] | 146 [141 to 161]
  TNF 365days | 153 [150 to 164] | 157 [151 to 167]
  IL10 90days | 155 [150 to 168] | 164 [160 to 173]
  IL10 365 days | 179 [168 to 188] | 182 [177 to 186]
  IL6 90days | 282 [224 to 334] | 349 [224 to 349]
  IL6 365days | 281 [223 to 418] | 262 [237 to 281]
  IL1 90days | 212 [194 to 234] | 215 [195 to 224]
  IL1 365days | 228 [209 to 258] | 228 [226 to 242]
  VEGF 90days | 82 [67 to 107] | 70 [57 to 140]
  VEGF 365days | 84 [46 to 141] | 45 [33 to 58]
  FGF 90days | 39 [35 to 44] | 43 [37 to 48]
  FGF 365days | 30 [26 to 37] | 29 [23 to 31]
  CD106 90days | 43222 [33422 to 59960] | 28564 [9732 to 55116]
  CD106 365days | 18324 [12261 to 54026] | 19614 [11721 to 26523]
  CD54 90days | 1512 [746 to 2594] | 1293 [666 to 4206]
  CD54 365days | 696 [217 to 1321] | 1664 [1309 to 2319]
Statistical Analysis 1: Comparison: Tacrolimus vs Everolimus; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Evaluation of Renal Function
Description: Evaluation of renal function (serum creatinine) 90 days after transplant and 365 days after transplant.
Time Frame: 90 days after transplant and 365 days after transplant
Measure: Median (Inter-Quartile Range); unit: mg/dL
Groups:
- Tacrolimus: Kidney transplant patients with living donors starting with the use of tacrolimus, mycophenolate sodium and prednisone without induction.
- Everolimus: Kidney transplant patients with living donors starting with the use of tacrolimus, mycophenolate sodium and prednisone without induction, and converted for use of mycophenolate sodium, everolimus, and prednisone after 90 days of kidney transplantation.
Arm/Group | Tacrolimus | Everolimus
Number analyzed (Participants) | 10 | 12
mg/dL
  Cr 90days | 1.6 [1.2 to 1.7] | 1.3 [1.05 to 1.66]
  Cr 365days | 1.4 [1.22 to 1.65] | 1.4 [0.95 to 1.47]
Statistical Analysis 1: Comparison: Tacrolimus vs Everolimus; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected during the followup of the study, which was done until the last biopsy, 1 year after transplant.
Description: Because the access to patients and files by the PI were limited as previous explained, serious adverses events were considered all cause mortality, and graft failure. Other adverse event was biopsy acute rejection. Withdrawn of the study by patient option, or because everolimus serum level was not reached, was recorded but not considered a adverse event. Hospitalizations were not considered adverse events because sometimes it weren't recorded by the office, and not reported to the PI.
Groups:
- Tacrolimus: Kidney transplant patients starting taking tacrolimus, mycophenolate sodium and prednisone, and keeping it the whole study.
- Everolimus: Kidney transplant patients taking tacrolimus, mycophenolate sodium and prednisone, and whom switched tacrolimus to everolimus 90 days after renal transplantation. Therefore the patients were taking everolimus, mycophenolate sodium and prednisone since 90 days after the transplant, and kept this way during the whole study
Arm/Group | Tacrolimus | Everolimus
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 0/15 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus (N=15) | Everolimus (N=15)
graft failure (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus (N=15) | Everolimus (N=15)
biopsy proven acute rejection (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Principal Investigator was out of Santa Casa de Misericordia de Belo Horizonte in the periods august-2012 to september-2013, and after december-2014. Data was so restricted mainly to cytokine analysis, acute rejection, graft failure and mortality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No